CLINICAL TRIAL: NCT04669093
Title: Person by Situation Interaction: Matching Suggestions to Participants' Motivational Styles
Brief Title: Individual Differences in Placebo Analgesic Effects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Tor Wager, Principal Investigator, Trustees of Dartmouth College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 230138
Record Dates: First submitted 2020-11-16; First posted 2020-12-16 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: This is a within-participant design. Each participant will participate in two sessions. In both sessions, an over-the-counter hand cream will be applied to their skin, accompanied by a placebo suggestion that the cream is analgesic. In one session, the suggestion will match the participant's motivational style, and in the other session the suggestion will not match their motivational style. The order of sessions will be counterbalanced across participants. Each session will also include a control condition, in which participants will be told that the cream has no affect. The same over-the-counter hand cream will be used in all sessions.
Who Masked: Participant
Masking Description: Participants will not be aware of the type of suggestion (or the fact there are different types of suggestions) during the experiment. They will be debriefed upon the study's conclusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Experimental): All participants will participate in two sessions, one with a placebo suggestion that matches the participant's motivational style, and one with placebo suggestion that does not match their motivational style, in a pseudo-random order.
  Interventions: Behavioral: Placebo cream- "promotion" suggestion; Behavioral: Placebo cream- "prevention" suggestion
- Control (Experimental): Each session will also include a control phase, in which the same cream will be applied, and participants will be instructed that the cream has no analgesic effects.
  Interventions: Behavioral: Control cream

INTERVENTIONS:
Behavioral: Placebo cream- "promotion" suggestion — Over-the-counter hand cream will be applied to participants' skin, but they will be told that they are given a highly efficient topical analgesic cream. The suggestion will be based on a "promotion" approach (promoting good feelings).
  Arms: Placebo
Behavioral: Placebo cream- "prevention" suggestion — Over-the-counter hand cream will be applied to participants' skin, but they will be told that they are given a highly efficient topical analgesic cream. The suggestion will be based on a "prevention" approach (preventing pain).
  Arms: Placebo
Behavioral: Control cream — In a control condition, with the same cream as in the placebo interventions, participants will be instructed that the cream is a control cream with no effects.
  Arms: Control

SUMMARY:
This study examines the effects of placebo suggestions tailored to match or mismatch individual participants' motivational styles-an issue of person-situation 'fit' with important effects in public health settings, but which has been ignored in past research.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants
* Dominant promotion focus or dominant prevention focus (based on our screening)

Exclusion Criteria:

* Currently or recently suffered from chronic pain (based on screening)
* Cannot tolerate heat pain applied to the forearm, based on a calibration task at the beginning of the experiment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-09-30 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in subjective ratings of acute thermal pain | Measured repeatedly, immediately after thermal stimuli on the day of participation. Averaged and compared across interventions.
  Following each thermal stimulus, participants are asked to rate how painful it was, on a semi-circular computerized scale. Ratings are based on the angle (0-180), with higher angle representing higher pain ratings. We will average and compare the pain ratings within participant across interventions.
Changes in subjective ratings of pain expectations | Measured repeatedly, immediately before thermal stimuli on the day of participation. Averaged and compared across interventions.
  Before each thermal stimulus, participants are asked to rate how painful they expect the next stimulus to be, on a semi-circular computerized scale. Ratings are based on the angle (0-180), with higher angle representing higher expectations ratings. We will average and compare the expectation ratings within participant across interventions.

SECONDARY OUTCOMES:
Facial expressions | Immediate response measured during painful stimulation on the day of participation. Averaged and compared across interventions.
  We will obtain facial video recordings of participants with a video camera. We will analyze these data according to Facial Action Units (facial expressions) that are known to be related to pain, and compare them across interventions.
Thermal imaging of the face | Immediate response measured during painful stimulation on the day of participation. Averaged and compared across interventions.
  We will obtain thermal recordings of participant's face with an infrared camera, and compare the heat signature of the face (the temperature in different parts of the face) across interventions.
Changes in skin conductance response measured with a Biopac device | Immediate response measured during painful stimulation on the day of participation. Averaged and compared across interventions.
  Skin conductance will be measured. We will compare the skin conductance response to pain stimuli within participant across interventions.
Changes in heart rate measured with a Biopac device | Immediate response measured during painful stimulation on the day of participation. Averaged and compared across interventions.
  Heart rate will be measured. We will compare the heart rate in response to pain stimuli within participant across interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Tor D Wager, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data will be publicly shared via public online platforms such as the Open Science Framework (OSF) and Github, and the NIMH Data Archive (NDA), according to the terms and conditions outlined on their website (https://ndar.nih.gov/contribute_data_sharing_regimen.html). Identifying information will not be released, including the facial videos, of which only non-identifiable features will be extracted and shared.
Time Frame: All data will be de-identified prior to sharing. Raw data will be submitted to NDA within one year from the end of data collection or 6 months from the acceptance date of the first primary study manuscript on the full dataset (excluding methods development papers), whichever is later. Analyzed data/maps of statistical results and models accompanying each paper will be submitted to NDA/OpenFMRI when the primary study manuscript is accepted.
Access Criteria: These data would generally be made available to any qualified investigator for neuroimaging studies only including:
  i. Research on any brain phenomenon; ii. Neuroimaging research on non-disease traits (intelligence, behavioral traits); iii. Methods development research.
  The requesting investigator must provide documentation of local IRB approval.
  These data would not be made available to:
  i. Any criminal justice organization, because data may not be used for any criminal justice applications; ii. Any commercial entity, because use of the data is limited to not-for-profit organizations and data may not be used for any commercial purposes.

DOCUMENTS (1):
  • Informed Consent Form (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT04669093/ICF_000.pdf